CLINICAL TRIAL: NCT00324675
Title: Effects of Rosiglitazone on Renal Hemodynamics and Proteinuria of Type 2 Diabetic Patients With Renal Insufficiency Due to Overt Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DN 2
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Type 2 Diabetes; Overt Diabetic Nephropathy
Keywords: type 2 diabetes,; glomerular filtration rate,; renal plasma flow,; endothelial dysfunction,; proteinuria,; diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria; Diabetic Nephropathies | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosiglitazone (Active Comparator)
  Interventions: Drug: Rosiglitazone
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — 4 mg tablets, bid, 12 months
  Arms: Rosiglitazone
Drug: Placebo — 2 tablets per day
  Arms: placebo

SUMMARY:
Objective:

To evaluate how rosiglitazone does influence the renal plasma flow, the glomerular filtration rate and the degree of proteinuria in type 2 diabetic patients with renal insufficiency due to overt diabetic nephropathy.

Background:

Diabetic nephropathy is a world wide public health concern of increasing proportions. It has become the most common single cause of end-stage renal disease in the United States and in Europe. Previous studies have already found agents modifying the renin-angiotensin-system (ACE inhibitors and angiotensin receptor blocker) to retard diabetic nephropathy. These agents are likely to exert multiple effects in the kidney. One of them appear to be their known ability to improve endothelial function and to change renal glomerular hemodynamics.

In a previous study we demonstrated an improvement of renal endothelial dysfunction in type 2 diabetic patients without end organ damage after treatment with rosiglitazone. In that study, rosiglitazone significantly reduced glomerular hyperfiltration. This was associated with a reduction of urinary albumin excretion. The observed effects are potentially important in the context of renal protection, provided that a similar beneficial effect of rosiglitazone is demonstrable in overt diabetic nephropathy (renal insufficiency, hypertension, proteinuria).

Hypothesis Rosiglitazone decreases proteinuria and improves renal hemodynamic function in patients with chronic renal insufficiency due to overt diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

type 2 diabetes mellitus -age between 40 and 75 years -well controlled HbA1c (< 7.5%) -chronic renal failure (creatinin clearance between 70 and 30 mL/(min x 1.73 m²) according to the Cockroft equation) -proteinuria > 300 mg / 24 hours

Exclusion Criteria:

type 1 diabetes -poorly controlled type 2 diabetes (HbA1c > 7.5%) or unstable blood glucose during the day (capillary blood glucose self monitoring) -elevation of ALT, AST or GGT more than 2.5 fold the upper normal value -CHF (more than grade 1 of NYHA) -uncontrolled hypertension -malignant tumorous disorder -hyper- or hypothyroidism -pregnant women -nursing women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pistrosch, M.D., Principal Investigator — Nephrology, Department of Medicine, University hospital Dresden
Locations (1):
- University hospital Dresden, Dresden, Germany

REFERENCES:
- [Derived] Pistrosch F, Passauer J, Herbrig K, Schwanebeck U, Gross P, Bornstein SR. Effect of thiazolidinedione treatment on proteinuria and renal hemodynamic in type 2 diabetic patients with overt nephropathy. Horm Metab Res. 2012 Nov;44(12):914-8. doi: 10.1055/s-0032-1314836. Epub 2012 Jun 21. PMID 22723267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment at medical clinic and outpatient department
Pre-assignment Details: 2 enrolled patients were excluded: one withdrew infromed consent, one developed anaphylactic reaction to sinistrin (used for renal function test)
Period: Overall Study
Arm/Group | Rosiglitazone | Placebo
Started | 14 | 14
Completed | 13 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 8 | 9 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.6) | 66.5 (8.5) | 66.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Germany | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Proteinuria
Time Frame: at baseline and after 6 and 12 mo of treatment
Population: per protocol
Measure: Mean (Standard Error); unit: g/24hr
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 13 | 14
g/24hr
  baseline | 2.4 (1.1) | 1.6 (0.6)
  6 mo | 1.2 (0.6) | 1.6 (0.8)
  12 mo | 1.5 (0.7) | 1.7 (0.8)

2. Secondary Outcome: Renal Hemodynamic
Time Frame: at baseline and after 6 and 12 mo of tretament
Reporting Status: Not Posted

3. Secondary Outcome: Renal Function
Time Frame: at abseline and after 6 and 12 mo
Reporting Status: Not Posted

4. Secondary Outcome: Adverse Event
Time Frame: every month or at occurence
Reporting Status: Not Posted

5. Secondary Outcome: HbA1c
Time Frame: at baseline and after 6 and 12 mo
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/14 | 2/14
Other Adverse Events (participants affected / at risk) | 12/14 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone (N=14) | Placebo (N=14)
sleep apnoe (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
atrial fibrillation with congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone (N=14) | Placebo (N=14)
peripheral edema (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
anemia new or worsening (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
hypoglycemia (Endocrine disorders) | 2 (2) | 0 (0)
painful calf or foot (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
hypotension (Vascular disorders) | 2 (2) | 0 (0)
common cold (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No